CLINICAL TRIAL: NCT04466904
Title: A Multiple Dose Human Tolerability and Pharmacokinetic Study of IBI362 in Chinese Patients With Type 2 Diabetes Mellitus and Poor Glycemic Control
Brief Title: Multiple-dose Tolerability and Pharmacokinetic of IBI362 in Chinese Patients With T2DM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362A101
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mazdutide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI362 low dose cohort (Experimental): Participants receive low dose level of IBI362, matched placebo or Dulaglutide administrated by multiple subcutaneous injection.
  Interventions: Drug: IBI362; Drug: Placebo; Drug: Dulaglutide
- IBI362 medium dose cohort (Experimental): Participants receive medium dose level of IBI362, matched placebo or Dulaglutide administrated by multiple subcutaneous injection
  Interventions: Drug: IBI362; Drug: Placebo; Drug: Dulaglutide
- IBI362 high dose cohort (Experimental): Participants receive high dose level of IBI362, matched placebo or Dulaglutide administrated by multiple subcutaneous injection
  Interventions: Drug: IBI362; Drug: Placebo; Drug: Dulaglutide

INTERVENTIONS:
Drug: IBI362 — Administrated by subcutaneous injection
Drug: Placebo — Administrated by subcutaneous injection
Drug: Dulaglutide — Administrated by subcutaneous injection

SUMMARY:
This trial is aimed to investigate the safety, tolerability, PK and PD of multiple subcutaneous injections of IBI362 in Chinese patients with type 2 diabetes who have poor glycemic control after lifestyle or metformin intervention

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial, the first trial to assess the safety, tolerability, and PK/PD of IBI362 administered as multiple injections in Chinese patients with type 2 diabetes. The investigators and subjects will be blinded to the study drug IBI362 and placebo. Dulaglutide will be used as an open-label active control group. In this trial, 42 eligible patients will be recruited and randomly allocated to three cohorts. Each corhot will be randomized as an 8:4:2 ratio to IBI362 (n = 8), placebo (n = 4), and Dulaglutide 1.5 mg (n = 2).

ELIGIBILITY:
* Eligibility Criteria： Inclusion Criiteria:

1. Male or female 18 to 75 years of age at the time of consent.
2. T2D patients with poorly controlled blood glucose treated with lifestyle intervention or stable dose of metformin (≥ 1000mg/day or maximum tolerated dose) within 2 months prior to screening.
3. HbA1c 7.5% ≤ 11.0% by local laboratory at screening.
4. Body mass index 20 ≤ BMI ≤ 35 kg/m2.

Exclusion Criteria:

1. Type 1 diabetes, special types of diabetes, or gestational diabetes.
2. Ketoacidosis or lactic acidosis within 6 months prior to screening.
3. History of severe hypoglycaemic episodes within 6 months prior to screening.
4. Acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, coronary intervention (except diagnostic angiography), transient ischemic attack (TIA), cerebrovascular accident, acute and chronic heart failure within 6 months before screening.
5. Clinically symptomatic liver disease, acute or chronic hepatitis, or transaminases (ALT and AST) and alkaline phosphatase (ALP) > 2 times the upper limit of normal and total bilirubin above the upper limit of normal at screening.
6. The patient was previously diagnosed with autonomic neuropathy, manifested as urinary retention, resting tachycardia, orthostatic hypotension and diabetic diarrhea.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
To assess the number and incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of IBI362 compared with placebo | From the first dose of study drug to week 19
  Number of subjects with treatment emergent adverse events and serious adverse events through the end of the follow-up period

SECONDARY OUTCOMES:
The PK/PD parameters of IBI362 in patients with T2DM | From Baseline to week 12
Evaluate the Peak Plasma Concentration (Cmax) of IBI362 in patients with T2DM | From Baseline to week 12
Evaluate the Area under the plasma concentration versus time curve (AUC) of IBI362 in patients with T2DM | From Baseline to week 12
Evaluate the Fasting Blood Glucose (FBG ) of IBI362 in patients with T2DM | From Baseline to week 12
Evaluate the Glucagon of IBI362 in patients with T2DM | From Baseline to week 12
Evaluate the Insulin of IBI362 in patients with T2DM | From Baseline to week 12
Evaluate the C-peptide of IBI362 in patients with T2DM | From Baseline to week 12
Number of Participants With Anti-IBI362 Antibodies | From the first dose of study drug to week 19
  Serum samples will be analyzed by an electrochemiluminescence (ECL)-based immunoassay for anti-IBI362 binding antibodies. Positive samples will be subsequently tested in a receptor-ligand binding bioassay for anti-IBI362 neutralizing antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- China Japan Friendship Hospital, Beijing, China

REFERENCES:
- [Derived] Jiang H, Pang S, Zhang Y, Yu T, Liu M, Deng H, Li L, Feng L, Song B, Han-Zhang H, Ma Q, Qian L, Yang W. A phase 1b randomised controlled trial of a glucagon-like peptide-1 and glucagon receptor dual agonist IBI362 (LY3305677) in Chinese patients with type 2 diabetes. Nat Commun. 2022 Jun 24;13(1):3613. doi: 10.1038/s41467-022-31328-x. PMID 35750681